CLINICAL TRIAL: NCT06056167
Title: The Efficacy and Safety of Degludec Insulin Use for Glycemic Control in Critically Ill Patients: A Prospective Interventional Study (Protocol)
Brief Title: Degludec Insulin Use in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Zainab Alduhailib, Consultant Critical Care Medicine, King Faisal Specialist Hospital & Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KingFaisal
Record Dates: First submitted 2023-09-13; First posted 2023-09-28 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus; Critical Illness; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Critical Illness; Hyperglycemia | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Degludec (Experimental)
  Interventions: Drug: Degludec insulin

INTERVENTIONS:
Drug: Degludec insulin — Enrolled patients will be initiated on regular insulin sliding scale (ISS) every 6 hours, administrated subcutaneously at 0600, 1200, 1800 and 2400 in patients who are nil per os and on intravenous fluid or parenteral nutrition or continuous tube feeding, according to King Faisal Specialist Hospital & Research Center (KFSH&RC) protocol.
  Patients with two capillary point of care glucose levels of > 10 mmol/L (180 mg/dl) will be initiated on insulin degludec at dose of 0.2 units/ kg.
  Dose adjustments will be carried out on daily basis based on blood glucose levels following a written protocol.

SUMMARY:
Background:

Dysglycemia in critically ill patients is common, where 40% to 54% of patients were found to be hyperglycemic on intensive care unit admission. Several randomized controlled trials (RCT) were conducted to address the importance of glycemic control during critical illness on patient's outcomes.

The American association of diabetes recommends initiation of insulin infusion for critically ill patients aiming to target glucose levels 140-180 mg/dl. However, several limitations prevent the use of insulin infusion in critically ill such as the requirements of frequent blood glucose measurement and nursing staff workload, which in turn led to the use of the subcutaneous rapid acting and basal insulin during critical illness. The evidence on the use of subcutaneous insulin therapy compared to insulin infusion is mainly derived from observational studies that showed conflicting results.

Multiple RCTs demonstrated the comparable efficacy of degludec versus glargine in blood glycemic control and better safety profile in terms of nocturnal hypoglycemia and severe hypoglycemia in the outpatient/inpatient diabetic population. Studies addressing the role, safety, and efficacy of degludec in critically ill patients are lacking.

Study aim:

To assess the effectiveness of using insulin degludec as basal insulin in conjunction with subcutaneous regular insulin sliding scale (ISS) in the glycemic control in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Newly admitted critically ill patients with diabetes and expected ICU stay ≥ 48 hours
* Medical or surgical ICU patients

Exclusion Criteria:

* Patients who were already started on insulin infusion based on physician discretion.
* Postoperative patients with expected ICU stay less than 48 hours
* Diabetic ketoacidosis or hyperosmolar hyperglycemic state.
* Patients with Do-Not-Attempt-Resuscitation (DNAR) status or imminent plan to palliation due to terminal disease.
* Refusal of the treating physician to enroll the patient into the study.
* Patients with diabetes mellitus Type 1.
* Patients who already eating prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The percentage of blood glucose readings at the target glycemic control 140- 180 mg/dL (7.8 -10 mmol/L). | until stopping the intervention and up to 28 days

SECONDARY OUTCOMES:
The average or mean blood glucose in the whole cohort | until stopping the intervention and up to 28 days
The proportions of patients achieving the target glycemic control | until stopping the intervention and up to 28 days
The time-spent at the target glycemic control 140- 180 mg/dL (7.8 -10 mmol/L). | until stopping the intervention and up to 28 days
The rate of developing hypoglycemia during therapy | until stopping the intervention and up to 28 days
Glucose variability during therapy | until stopping the intervention and up to 28 days
To determine the covariates associated with failure to achieve target glycemic control | During therapy and up to 28 days
  To assess the factors that are associated with failure to achieve the target glycemic control (using regression analysis).
To determine the covariates associated with the development of hypoglycemia | During therapy and up to 28 days
  To assess the factors that are associated with the development of hypoglycemia (using regression analysis).
The rate of 28-day Mortality | Censored at day 28
  Death rate at day 28
Intensive care unit (ICU) length of stay | Censored at day 28

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes